CLINICAL TRIAL: NCT04068454
Title: The Use of Virtual Reality in Shoulder Reeducation : Interests and Limits.
Brief Title: Virtual Reality in Reeducation : Application to Shoulder Affections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2019-03-21; First posted 2019-08-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Scapular Dyskinesis; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical rehabilitation group (Active Comparator)
  Interventions: Other: EBM rehabilitation exercises
- virtual reality group (Experimental)
  Interventions: Device: Virtual reality device

INTERVENTIONS:
Device: Virtual reality device — Functional exercises will be done by virtual reality group
  Arms: virtual reality group
Other: EBM rehabilitation exercises — scapular exercises will be done
  Arms: classical rehabilitation group

SUMMARY:
The objective of this study is to assess the interest and the efficiency of virtual reality in functional rehabilitation of shoulder pain and shoulder injuries. Participants will follow a 12-week rehabilitation program based either on exercises or on a program integrating virtual reality. Results obtained with classical rehabilitation will be compared with the one obtained virtual reality.

DETAILED DESCRIPTION:
Fifty people will be included in the study. Then, they were randomly separated in two groups : 25 people will do the "classical rehabilitation" and the other 25 will have a treatment with virtual reality.

Each group (virtual reality and "classical rehabilitation") is going to follow 12 weeks of rehabilitation, at a rate of 2x 30 minutes per week. In "virtual reality group", each session will be divided in two parts : 15 minutes of virtual reality exercises and 15 minutes of exercises from "classical program". Exercises suggested in the classical program have been chosen among evidence based exercises described in literature.

Before the beginning of rehabilitation sessions, participants will be assessed at the Laboratory of Human Motion Analysis of the University of Liege. At this place, EMG activity of periscapular muscles (upper trapezius, lower trapezius and serratus anterior) (Delsys Trigno) , 3D scapular kinematics (Codamotion) will be assessed on the painful side when doing shoulder elevations in sagittal and in frontal planes. Maximum isometric strength will also be assessed using handheld dynamometer (MicroFet2) in 3 different positions (SeatedU90°, SeatedU125°, Prone-v-thumbs up)

This first evaluation will be done after the 12 week of rehabilitation too, with the same method.

Participants will also have to complete Dash (Disability of the Arm, Shoulder and Hand) questionnaire 3 times during the study (at the beginning, at 6 weeks and at the end of the study). Moreover, pain score will be asked to participants at each rehabilitation session.

ELIGIBILITY:
Inclusion criteria:

* unilateral scapular dyskinesis
* positive scapular assistance test and positive resistance test
* shoulder pain
* ability to play sport despite shoulder pain
* one or more positive tendinous tests

Exclusion criteria :

* traumatic history of shoulder injury in the last 6 months
* surgical history at shoulder or cervical location
* scoliosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Score of Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | change from baseline at 12 weeks
  Functional ability and quality of life will be assessed using this questionnaire, with a maximal score of 100

SECONDARY OUTCOMES:
Shoulder pain | change from baseline at 12 weeks
  Shoulder pain will be assessed, with a maximum score of 10 (0= no pain and 10= maximum pain)
EMG activity | Change from baseline at 12 weeks
  EMG activity of upper trapezius, lower trapezius and serratus anterior will be assessed using surface EMG
3D scapular motion | Change from baseline at 12 weeks
  Scapular motion will be assessed when doing elevations in sagittal and frontal planes (in loaded and unloaded conditions)
Maximum voluntary isometric contraction | Change from baseline at 12 weeks
  Maximum isometric strength will be assessed in 3 different positions (SeatedU90°, SeatedU125°, Prone-v-thumbs up) with handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Camille Tooth, Principal Investigator — University of Liege
Locations (1):
- University of Liege, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No